CLINICAL TRIAL: NCT00745199
Title: Phase II Study of the Effect of Oral Cromolyn Sodium on Uremic Pruritus and Serum Tryptase Levels of Hemodialysed Patients
Brief Title: Evaluating the Effect of Cromolyn Sodium in Uremic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Dr.Ghazal Vessal PharmD, BCPS, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4146
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: End Stage Renal Disease; Pruritus
Keywords: End Stage Renal Disease; Cromolyn Sodium; Pruritus; Tryptase
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Patients on hemodialysis with pruritus, receiving cromolyn sodium
  Interventions: Drug: cromolyn sodium
- 2 (Experimental): patients on hemodialysis with pruritus, receiving placebo
  Interventions: Drug: placebo
- 3 (No Intervention): Patients on hemodialysis but without pruritus who do not receive any treatment.

INTERVENTIONS:
Drug: cromolyn sodium — oral cromolyn sodium, capsule 135mg, 1 capsule 3 times daily for 8 weeks
  Arms: 1
Drug: placebo — capsule contains 135 mg lactose, 1 capsule 3 times daily for 8 weeks
  Arms: 2

SUMMARY:
Pruritus is a major disorder among the skin derangements in advanced renal failure. Recent information suggests that interactions between dermal mast cells and distal ends of nonmyelinated C fibers may be important in the precipitation and regulation of the sensory stimuli.Patients having uremic pruritus have been noted to have increased levels of plasma histamine and tryptase as well as increased numbers of dermal mast cells.Cromolyn sodium is a mast cell stabilizing agent that inhibits degranulation of mast cells and the release of histamine, tryptase, and leukotrienes. It is hypothesized that oral cromolyn sodium may attenuate uremic pruritus by decreasing serum tryptase level.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients > 18 yo suffering from pruritus for at least 6 weeks, and who have not responded to other drugs
* Willing and able to give informed concent

Exclusion Criteria:

* Known dermatologic, liver, metabolic disease, or any other disease or condition other than ESRD that causes pruritus
* Lactase deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
pruritus | 3 months

SECONDARY OUTCOMES:
serum tryptase level | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghazal Vessal, PharmD, BCPS, Study Director — Shiraz University of Medical Sciences; Mohammad Mahdi Sagheb, MD, Principal Investigator — Shiraz University of Medical Sciences; Saman Shilian, Pharm student, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical sciences, Nemazi and Faghihi Hospital, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264